CLINICAL TRIAL: NCT07012733
Title: A Randomized Controlled Trial Comparing the Effects of Thoracic Mobilization and Conventional Respiratory Therapy on Cough Capacity, Dyspnea, and Pulmonary Function in Patients With Restrictive Lung Disease
Brief Title: Thoracic Mobilization for Restrictive Lung Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chungnam National University Sejong Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNUSH2025-04-001; CNUSH2025-04-001 (Other: Chungnam National University Sejong Hospital)
Record Dates: First submitted 2025-05-22; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Restrictive Lung Disease
Keywords: thoracic mobilization; pulmonary function; cough capacity; dyspnea; restrictive pulmonary disorder
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-group clinical trial comparing thoracic mobilization techniques to conventional respiratory therapy in patients with restrictive lung disease.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to group assignment to minimize detection bias during post-intervention evaluations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic mobilization group (Experimental): Participants receive thoracic mobilization techniques
  Interventions: Other: Thoracic mobilization; Other: conventional therapy
- conventional therapy group (Active Comparator): Participants receive conventional respiratory therapy
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: Thoracic mobilization — Participants in this group will receive thoracic mobilization techniques in addition to conventional respiratory therapy. Thoracic mobilization will be delivered by a licensed physical therapist using passive manual techniques targeting the thoracic spine and rib cage to improve chest wall mobility and respiratory function.
  Arms: Thoracic mobilization group
Other: conventional therapy — Participants in this group will receive conventional respiratory therapy, including diaphragmatic breathing, pursed-lip breathing, and chest expansion exercises. The therapy will be administered by a licensed physical therapist following standard pulmonary rehabilitation protocols.

SUMMARY:
This study aims to investigate the immediate effects of thoracic mobilization techniques on cough capacity, dyspnea, and pulmonary function in patients with restrictive lung disease. The intervention will be applied in a single session, and outcomes will be measured before and after the intervention to evaluate short-term physiological changes.

DETAILED DESCRIPTION:
Restrictive lung disease (RLD) is characterized by reduced lung compliance and limited thoracic mobility, leading to decreased lung volume and impaired respiratory function. Manual therapy interventions such as thoracic mobilization have been proposed to improve chest wall flexibility and enhance respiratory efficiency. However, few studies have examined the immediate clinical effects of such interventions in RLD patients.

This single-group pre-post interventional study will evaluate the short-term outcomes of thoracic mobilization techniques on cough capacity (as measured by peak cough flow), dyspnea (via Borg scale), and pulmonary function (forced vital capacity [FVC], forced expiratory volume in 1 second [FEV1]). The results are expected to provide preliminary evidence on the effectiveness of thoracic mobilization for improving respiratory performance in individuals with RLD.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older
* Currently receiving respiratory therapy at C Hospital in Sejong City
* Pulmonary function test indicating restrictive pattern: FVC < 80% and FEV1/FVC ≥ 70%
* FVC above the lower limit of normal (LLN) for age and sex
* Diagnosed with restrictive lung disease, such as idiopathic pulmonary fibrosis, scoliosis, or neuromuscular disorders (e.g., myopathy, amyotrophic lateral sclerosis)

Exclusion Criteria:

* FEV1/FVC ratio < 70%
* Evidence of airway obstruction on pulmonary function testing

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-09 (Estimated); Primary Completion 2025-11-18 (Estimated); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function test | Immediately before and immediately after intervention on Day 1
  Pulmonary function will be assessed using a standard spirometry test, including FVC and FEV1. The test will be conducted by a trained technician according to ATS/ERS guidelines to evaluate respiratory function.

SECONDARY OUTCOMES:
Cough peak flow | Immediately before and immediately after intervention on Day 1
  Cough peak flow will be measured using a peak flow meter. Participants will be instructed to perform a maximal voluntary cough following a deep inspiration, and the highest value from three trials will be recorded. The assessment will be conducted by a trained therapist to evaluate cough capacity.
Dyspnea | Immediately before and immediately after intervention on Day 1
  Dyspnea will be assessed using the modified Borg scale, a subjective rating scale ranging from 0 (no breathlessness) to 10 (maximum breathlessness). Participants will rate their perceived level of dyspnea at rest following the intervention. The assessment will be administered by a trained therapist.

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam National University Sejong Hospital, Sejong, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared upon reasonable request for academic purposes. Data will be available from 6 months after publication of the primary results for a period of 2 years.
Supporting Information: Study Protocol, SAP
Time Frame: IPD and supporting documents will be available beginning 6 months after publication of the primary results and will be accessible for up to 2 years.
Access Criteria: De-identified individual participant data and supporting documents will be available to qualified researchers for academic purposes. Requests must include a methodologically sound proposal and will be subject to approval by the study team. Data will be shared through secure institutional data transfer.

REFERENCES:
- [Background] Kelzuyuki, T., Noriko, S. The immediate effect of chest mobilization tech. in patients of COPD. The Journal of Japanese Physical Therapy Association.(JPTA). 2007;34(2): 20070420.